CLINICAL TRIAL: NCT05982106
Title: A Randomized, Open-label, Single-center, Two-cycle, Two-crossover Phase I Clinical Trial Evaluating the Effect of Food on the Pharmacokinetics of TQ05105 Tablets in Healthy Adult Subjects
Brief Title: To Evaluate the Effect of Food on the Pharmacokinetics of TQ05105 Tablets in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TQ05105-I-03
Record Dates: First submitted 2023-07-07; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ05105 Tablets (fasted) (Experimental): TQ05105 tablets was administered on fasted state in the first cycle for Group A and the second cycle for Group B.
  Interventions: Drug: TQ05105 Tablets
- TQ05105 Tablets (fed) (Experimental): TQ05105 tablets was administered on fed state in the second cycle for Group A and the first cycle for Group B.
  Interventions: Drug: TQ05105 Tablets

INTERVENTIONS:
Drug: TQ05105 Tablets — TQ05105 tablet is a novel JAK2 inhibitor.

SUMMARY:
TQ05105 is a class 1 new drug with a new chemical structure developed by Chia Tai Tianqing Pharmaceutical Group Co., Ltd. It is a Janus Kinase 2 （JAK2）inhibitor and can be used to treat JAK2 target-related diseases. This study is a randomized, open-label, single-center, two-cycle, two-crossover Phase I clinical trial evaluating the effect of food on the pharmacokinetics of TQ05105 tablets in healthy adult subjects. Pharmacokinetic effects and safety after oral administration of TQ05105 tablets.

ELIGIBILITY:
Inclusion Criteria:

* 1 Sign the informed consent form before the test, and fully understand the test content, process and possible adverse reactions;
* 2 Able to communicate well, understand and complete the research in accordance with the requirements of the experimental protocol;
* 3 Male and female subjects aged 18 to 65 (including 18 and 65 years old);
* 4 Body mass index (BMI) ≥ 18 and ≤ 28kg/m2, and male weight ≥ 50 kg and female weight ≥ 45 kg;
* 5 Health status: no history of heart, liver, kidney, digestive tract, nervous system, mental abnormalities and metabolic abnormalities, and physical examination showed normal or abnormal blood pressure, heart rate, electrocardiogram, respiratory system, liver, kidney function and blood picture without clinical significance;
* 6 The subjects have no pregnancy plans and voluntarily take effective contraceptive measures from 2 weeks before the administration to at least 6 months after the last use of the study drug.

Exclusion Criteria:

* 1 Patients with neuropsychiatric system, respiratory system, cardiovascular system, digestive tract system, blood-lymphatic system, liver and kidney insufficiency, endocrine system, musculoskeletal system disease or other diseases in the past, and the researcher judges that the past medical history may have an adverse effect on the drug. Metabolic or safety effects;
* 2 Those with allergic constitution or a history of two or more food or drug allergies in the past;
* 3 Those with multiple factors that affect oral drugs (such as inability to swallow, gastrointestinal diseases);
* 4 Taking any prescription, over-the-counter, vitamin product or herbal medicine within 1 month before taking the study drug;
* 5 Take CYP3A4 inhibitors or inducers within 1 month before screening or before study medication;
* 6 Those who have taken special diets (including grapefruit, etc.) or exercised vigorously within 14 days before screening, or have other factors that affect drug absorption, distribution, metabolism, and excretion;
* 7 aboratory examinations during the screening period are abnormal and have clinical significance;
* 8 Blood donation or massive blood loss (> 450mL) within 3 months before taking the study drug;
* 9 Participated in any drug clinical trial within 3 months before taking the study drug;
* 10 Smoking more than 5 cigarettes per day within 3 months before the test;
* 11 Positive breath test for alcohol or a history of alcohol abuse within 2 weeks before screening (drinking 14 units of alcohol per week: 1 unit = 360mL of beer or 45mL of spirits with an alcohol content of 40% or 150mL of wine);
* 12 Those who are positive for drug screening or have used drugs in the 3 months before the test;
* 13 Inability to tolerate venipuncture for blood collection or poor vascular condition;
* 14 Subjects have a history of herpes zoster within 1 month before screening;
* 15 The subject is unable to complete the trial due to personal reasons;
* 16 Other investigators deem it unsuitable for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Area under the drug-time curve (AUC) | 1 hour before administration and 10, 20, 30, 45 minuets, 1, 1.5, 2, 2.5, 3 ,3.5, 4, 6, 8, 12, 24 hours after administration
  Area under the drug-time curve
Maximum Concentration (Cmax) | 1 hour before administration and 10, 20, 30, 45 minuets, 1, 1.5, 2, 2.5, 3 ,3.5, 4, 6, 8, 12, 24 hours after administration
  Maximum concentration

SECONDARY OUTCOMES:
Time to maximum concentration following drug administration (Tmax) | 1 hour before administration and 10, 20, 30, 45 minuets, 1, 1.5, 2, 2.5, 3 ,3.5, 4, 6, 8, 12, 24 hours after administration
  Time to maximum concentration following drug administration
Apparent terminal elimination half-life following drug administration (t1/2) | 1 hour before administration and 10, 20, 30, 45 minuets, 1, 1.5, 2, 2.5, 3 ,3.5, 4, 6, 8, 12, 24 hours after administration
  Apparent terminal elimination half-life following drug administration
Apparent volume of distribution (Vd/F) | 1 hour before administration and 10, 20, 30, 45 minuets, 1, 1.5, 2, 2.5, 3 ,3.5, 4, 6, 8, 12, 24 hours after administration
  Apparent volume of distribution
Clearance rate (CL/F) | 1 hour before administration and 10, 20, 30, 45 minuets, 1, 1.5, 2, 2.5, 3 ,3.5, 4, 6, 8, 12, 24 hours after administration
  Clearance rate
Adverse event rate | Baseline up to 24 hours after administration
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Body temperature | 1 hour before administration and 1, 4, 12, 24 hours after administration
  Monitor the safety indicators of subjects during the trial
Pulse | 1 hour before administration and 1, 4, 12, 24 hours after administration
  Monitor the safety indicators of subjects during the trial
Blood pressure | 1 hour before administration and 1, 4, 12, 24 hours after administration
  Monitor the safety indicators of subjects during the trial

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China

REFERENCES:
- [Derived] Dai J, Cheng Y, Zhou Y, Wang Y, Liu Z, Ren Q, Su Z, Deng Q, Yang H, Cui Y. Food effect trial of the pharmacokinetics and safety of TQ05105 in healthy Chinese subjects. Cancer Chemother Pharmacol. 2025 Feb 10;95(1):31. doi: 10.1007/s00280-025-04754-z. PMID 39924599